CLINICAL TRIAL: NCT05074641
Title: Comparison Of Direct Myofascial Release And Bowen's Technique For Non-Specific Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC-00942 Shahzana khalid
Record Dates: First submitted 2021-09-29; First posted 2021-10-12 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-02

CONDITIONS: Neck Pain
Keywords: Pain; Range of motion; Myofascial release; Bowen therapy; Anxiety
MeSH Terms: conditions — Neck Pain; Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct myofascial release treatment (Experimental): Myofascial Release will be applied with Forearm and/or ulnar border of the palm. Deep Pressure will be applied and glided medially towards the base of the neck and/ or towards the upper scapular region
  Interventions: Other: Direct myofascial release treatment
- Bowen therapy (Active Comparator): Thumb of the therapist will be placed on the top of the targeted muscle. The skin will be carried away gently from the spine without disturbing the muscle. The thumb was then hooked into the lateral aspect of the muscle to form a pressure on the muscle. Then the thumb will be flattened in the medial direction, when this happened the muscle would plop or respond in some way.
  Interventions: Other: Bowen therapy

INTERVENTIONS:
Other: Direct myofascial release treatment — Myofascial Release will be applied with Forearm and/or ulnar border of the palm. Deep Pressure will be applied and glided medially towards the base of the neck and/ or towards the upper scapular region
  Arms: Direct myofascial release treatment
Other: Bowen therapy — Thumb of the therapist will be placed on the top of the targeted muscle. The skin will be carried away gently from the spine without disturbing the muscle. The thumb was then hooked into the lateral aspect of the muscle to form a pressure on the muscle. Then the thumb will be flattened in the medial direction, when this happened the muscle would plop or respond in some way.
  Arms: Bowen therapy

SUMMARY:
Neck pain is described as pain in the neck region that may or may not radiate to both the upper limbs and that will last for at least one day. Non-specific neck pain is the common cause of neck symptoms that is mainly due to mechanical causes, postural problem, depression, anxiety or occupational activities. Poor posture causes abnormal muscle loading and muscle injury

DETAILED DESCRIPTION:
Neck pain is described as pain in the neck region that may or may not radiate to both the upper limbs and that will last for at least one day.Poor posture causes abnormal muscle loading and muscle injury.It becomes a constant source of neck pain and instability. It reduces range of motion and weakens the shoulder and neck muscles. According to a population based survey the prevalence of lifetime neck pain ranges from 67% to 87%.

Trigger points cause myofascial pain syndrome which is among the leading cause of non-specific neck pain. Myofascial release technique (MRT) is often used to treat non-specific neck pain.Another therapy that focuses on myofascial work is Bowen therapy that follows a dynamic approach to release fascia and muscles. The technique involves very gentle cross fiber movements that are applied on fascia, muscles, tendons and viscera to induce the effect. The technique is applied at specific body regions following specific sequences with regular rest intervals that cause fascial stretching. The technique consists of slightly picking up muscles and then rolling the muscles to direct them toward a specific region of body. The rest periods help the body to integrate and absorb the effects of therapy. The sensory impulses caused by the Bowen therapy interact with nervous system and realign and correct the disturbed mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Chronic non-specific neck pain ≥ 3 months without symptoms radiating to the upper limbs
* Presence of a maximum of 1-2 active Myofascial Trigger Points
* Pain of more than 3 on a NPRS
* For the diagnosis of a Trigger Point, compliance with the following criteria:

  * (1) A hypersensitive spot in a palpable taut band,
  * (2) Palpable or visible local twitch on pincer palpation
  * (3) Reproduction of referred pain elicited by palpation of the sensitive spot.

Exclusion Criteria:

* Diagnosed with cervical radiculopathy or myelopathy
* Neck Pain due to trauma, fractures, or whiplash; neoplasia, severe osteoporosis, infectious, or inflammatory processes;
* Patients with pacemakers, congenital anomalies, previous neck surgery
* Patients diagnosed with fibromyalgia syndrome according to the American College of Rheumatology criteria

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale | for two weeks
  The Numeric pain rating scale is an 11-point numeric scale, it is the segmented numeric version of the visual analog scale. Subjects will be asked to mark/select a whole number for 0-10 that best describes their perceived pain intensity of the last 24 hours. zero indicates no pain and 10 is worst possible pain. assessment to be done at base line and after 2 weeks
Goniometer for Cervical Range of Motion | for two weeks
  The active cervical range of motion (CROM) will be measured in sitting posture by using a universal goniometer, which consists of two arms; one that is stationary and one that is moveable. assessment to be done at base line and after 2 weeks
Neck Disability Index | for two weeks
  it is a 10-item self-report questionnaire that measures the patient's disability related to his/her neck pain. It is the most commonly used questionnaire for neck disability; its reliability and validity has been demonstrated in many literatures and languages.its minimum score is zero no disability and 50 is maximum disability. Assessment to be done at base line and after 2 weeks
Depression Anxiety Stress Scale (DASS) | for two weeks
  DASS is a reliable and validated tool commonly administered to measure the level of stress, depression and anxiety of the respondent. It is 42-item questionnaire that focuses on low mood, motivation, self-esteem, physiological arousal, perceived panic, fear, tension and irritability. Respondent answer each question by indicating the extent on a 4-point scale. In this study Urdu version of DASS is used which has concurrent validity of .87 for normal subjects and .84 for clinical population and .89 reliability. its minimum value is zero which is normal and maximum is 34 plus which is stress. Assessment to be done at base line and after 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Maria Khalid, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No